CLINICAL TRIAL: NCT05714683
Title: A Multi-centre, Prospective, Open-label, Single-arm, Non-interventional, Regulatory Post Marketing Surveillance (rPMS) Study of Rybelsus® (Oral Semaglutide) to Evaluate Safety and Effectiveness in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in Korea
Brief Title: Regulatory Post Marketing Surveillance (rPMS) Study of Rybelsus (Oral Semaglutide) to Evaluate Safety and Effectiveness in Patients With Type 2 Diabetes Mellitus in Routine Clinical Practice in Korea
Status: Not yet recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4652; U1111-1243-9500 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with T2DM: All participants will be treated with Rybelsus for 26 weeks according to routine clinical practice at the discretion of the treating physician according to the label approved by Ministry of Food and Drug Safety (MFDS).
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — All participants will be treated with oral semaglutide for 26 weeks according to routine clinical practice at the discretion of the treating physician according to the label approved by MFDS. The prescription of semaglutide will be separated from the decision to include the participant in the study.
  Other Names: Rybelsus

SUMMARY:
The aim of this study is to assess the safety and effectiveness of Rybelsus initiated according to label in adults with Type 2 Diabetes Mellitus (T2DM) under routine clinical practice conditions. Participants will get Rybelsus as prescribed by study doctor. The study will last for about 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The decision to initiate treatment with commercially available Rybelsus has been made by the participant/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
* The participant with T2DM is scheduled to start treatment with Rybelsus based on the clinical judgment of their treating physician as specified in the approved label in Korea
* Informed consent is obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study
* Male/female age greater than or equal to (>=) 19 years at the time of signing informed consent

Exclusion Criteria:

* Participants who are or have previously been on Rybelsus therapy
* Known or suspected hypersensitivity to Rybelsus, the active substance or any of the excipients
* Previous participation in this study. Participation is defined as having given informed consent in this study
* Female participant who is pregnant, breast-feeding or intends to become pregnant and is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by Korea regulation or practice)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Family or personal history of multiple Endocrine Neoplasia Type 2 (MEN 2) or Medullary Thyroid Carcinoma (MTC)

Min Age: 19 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult participants with T2DM, who initiate treatment with Rybelsus under routine clinical practice in Korea.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Number (Incidence) of adverse events (AEs) | From baseline (week 0) to 26 weeks
  Measured as count of events.

SECONDARY OUTCOMES:
Number (Incidence) of hypoglycaemia Level 3 or Level 2 | From baseline (week 0) to 26 weeks
  Hypoglycaemia Level 3 or Level 2 according to American Diabetes Association (ADA) guideline 2020 refers to: 1) Level 2: Glucose less than (<) 54 milligrams per deciliter (mg/dL) (3.0 millimoles per liter [mmol/L]); 2) Level 3: A severe event characterized by altered mental and/or physical status requiring assistance for treatment of hypoglycaemia. Measured as count of events.
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to 26 weeks
  Measured in percentage (%).
Participants achieving HbA1c target <7.0% | At 26 weeks
  Measured as count of participants (Yes/No).
Change in fasting blood glucose (FBG)/fasting plasma glucose (FPG) | From baseline (week 0) to 26 weeks
  Measured in mg/dL.
Change in post prandial blood glucose (PPBG)/post prandial plasma glucose (PPPG) | From baseline (week 0) to 26 weeks
  Measured in mg/dL.
Change in body weight | From baseline (week 0) to 26 weeks
  Measured in kilogram (kg).
Dose of Rybelsus | At 26 weeks
  Measured in milligrams per day (mg/day).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com